CLINICAL TRIAL: NCT07244536
Title: Health-related Quality of Life in Elderly Adults Following Physical Exercise and Cognitive Training: a Randomized-controlled Trial
Brief Title: Effects of Physical Exercise and Cognitive Training on Quality of Life in Elderly Adults
Acronym: HELIOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Fabio Manfredini, Full Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 416/2025/Sper/UniFe
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Elderly (People Aged 65 or More)
Keywords: elderly; exercise; cognitive training; quality of life
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Exercise Program + Cognitive training (Experimental): In addition to the exercise program, participants will be given a series of cognitive exercises aimed at improving prospective memory through the performance of certain oral tasks, administered by a member of the research team.
  All cognitive exercises will be adapted to the cognitive abilities of the participants.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Structured Exercise Program + Cognitive stimulus (Experimental): In addition to the exercise program, people will receive a short video lasting less than 10 minutes on their smartphone or tablet before the exercise session (or at home). At the end of the video, they will be asked to complete a 10-question questionnaire (also delivered via smartphone or tablet) with True or False answer options.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Structured Exercise Program (Active Comparator): The program includes 75-minute training sessions twice a week, for a total of 24 training sessions over 12 weeks. Each training session will be divided into a warm-up, training phase and cool-down, and will include aerobic exercises, resistance training, balance exercises, mobility exercises and stretching.
  The exercise program will be the same for all the three groups
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — The program includes 75-minute training sessions twice a week, for a total of 24 training sessions over 12 weeks. Each training session will be divided into a warm-up, training phase and cool-down, and will include aerobic exercises, resistance training, balance exercises, mobility exercises and stretching.
  Arms: Structured Exercise Program
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — In addition to the exercise program, Participants will be given a series of cognitive exercises aimed at improving prospective memory through the performance of certain oral tasks, administered by a member of the research team. All cognitive exercises will be adapted to the cognitive abilities of the participants.
  Arms: Structured Exercise Program + Cognitive stimulus
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — In addition to the exercise training, people will receive a short video lasting less than 10 minutes on their smartphone or tablet before the exercise session (or at home). At the end of the video, they will be asked to complete a 10-question questionnaire (also delivered via smartphone or tablet) with True or False answer options.
  Arms: Structured Exercise Program + Cognitive training

SUMMARY:
The aim of the study is to investigate the effectiveness of three different types of intervention, based on physical exercise and/or cognitive stimulation or training, on quality of life, cognition and mobility, on a population of older adults, who are most at risk of functional and cognitive decline

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age ≥ 70 years
* Provision of the informed consent form

Exclusion Criteria:

* Absolute contraindications to physical exercise (e.g. NYHA class IV heart failure, unstable angina, etc.)
* Pregnancy
* Severe cognitive impairment, defined as a MoCa score ≤ 12
* Severe visual impairment or blindness

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life assessed by the short-form 36 (SF-36) questionnaire | Baseline; end of the program (3-month); Follow-up (6-month)
  This is a generic questionnaire that contains 36 questions referring to 8 specific domains related to patient health over the previous 4 weeks. For each specific domain, the score ranges from 0 (lowest quality of life) to 100 (highest quality of life).

SECONDARY OUTCOMES:
Quality of life assessed by the Quality of Life in Alzheimer's Disease (QOL-AD) questionnaire | Baseline; end of the program (3-month); Follow-up (6-month)
  QOL-AD consists of 13 questions covering various aspects of daily life, such as physical health, energy, mood, relationships and the ability to enjoy enjoyable activities. The combined scores of the patient and caregiver provide a more comprehensive and accurate picture of the person's overall well-being. The scale has a score ranging from 13 (lowest quality of life) to 52 (highest quality of life).
Cognitive capacity assessed by the Montreal Cognitive Assessment (MoCA) | Baseline; end of the program (3-month); Follow-up (6-month)
  MoCA is a 30-point test evaluates cognitive function. Its primary purpose is to detect mild cognitive impairment (MCI). The score goes from 0 (maximal cognitive deficit) to 30 (normal cognitive function).
Executive function and processing speed assessed by the Trail Making Test (TMT) | Baseline; end of the program (3-month); Follow-up (6-month)
  TMT is neuropsychological test that assesses a person's cognitive function, specifically focusing on visual attention, processing speed, and executive function. The test consists of two parts, the score is based on the time it takes to complete each part, with shorter times indicating better performance.
Walking endurance assessed by the 6-Minute Walking Test (6MWT) | Baseline; end of the program (3-month); Follow-up (6-month)
  The patients will be instructed to walk back and forth on a 20-meter corridor aiming at covering as much distance as possible. The total distance covered (6MWD) will be measured in meters
Short Physical Performance Battery (SPPB) | Baseline; end of the program (3-month); Follow-up (6-month)
  It is a specific assessment for the elderly population, consisting of three functional tests that measure postural stability, the ability to walk safely, and lower limb muscle strength. Higher scores indicate better functional ability. The scale goes from 0 (lowest functional ability) to 12 (highest functional ability).
Manual grip strength using the Handgrip Test (HT) | Baseline; end of the program (3-month); Follow-up (6-month)
  The test is performed using a dynamometer: the subject grabs the handle of the device with maximum strength, and the maximum value of force expressed in kilograms is recorded.
Sleep quality through the Pittsburgh Sleep Quality Index (PSQI) | Baseline; end of the program (3-month); Follow-up (6-month)
  It refers to the last 30 days and analyses seven components. The total score ranges from 0 to 21. A score above 5 indicates poor sleep quality.
Timed Up-and-Go test | Baseline; end of the program (3-month); Follow-up (6-month)
  This test ask the participant to stand up from a standard chair, walk for three meters, turn around a cone and get back to the starting point and seating. The total timed elapsed will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Esercizio Vita, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided